CLINICAL TRIAL: NCT03411278
Title: Effect of Deep Oscillation Treatment as a Method for Recovery After Fatiguing Soccer Training. A Randomized Cross-Over Study
Brief Title: Effect of Deep Oscillation Treatment as a Method for Recovery in Soccer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: IMPDO1
Record Dates: First submitted 2018-01-18; First posted 2018-01-26 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Sports Physical Therapy
Keywords: recovery; deep oscillation; soccer; sports; training; electrotherapy; physical therapy
MeSH Terms: interventions — Electric Stimulation Therapy

STUDY DESIGN:
Intervention Model Description: A randomized, cross-over, repeated measures design is used to evaluate the effects of DO on recovery. At random in study phase I the half of the group performs a DO self-treatment twice daily (4 applications) for 15 minutes each, whereas the other half gets no intervention. After a washing out period in study phase II a crossover will be performed. The same protocol is performed again, whereas the other half of the participants carries out the DO intervention .
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Deep Oscillation (DO) self treatment (Experimental): DO self treatment with the device "mobile" (Physiomed, Laipersdorf, Germany; U.S. patent 7,343,203 B2). The device produces an alternating electrostatic field, which results in a low-frequency vibration penetrating the tissue. The Field is pulsed at a frequency of 90 Hz. For self-treatment, each volunteer is given an apparatus to take home. An applicator with a diameter of 9 cm is used. The treatment will be carried out in the morning and evening for 15 minutes each in supine position on a sofa. In accordance with the technique of classical manual lymphatic drainage, stroking and circular movements in the upper and lower leg and the inguinal area take place in a fixed order.
  Interventions: Device: Deep Oscillation (DO)
- No intervention, control (No Intervention): No intervention

INTERVENTIONS:
Device: Deep Oscillation (DO) — DO self treatment with the device "mobile" (Physiomed, Laipersdorf, Germany; U.S. patent 7,343,203 B2).The device produces an alternating electrostatic field, which results in a low-frequency vibration penetrating the tissue. The Field is pulsed at a frequency of 90 Hz. For self-treatment, each volunteer is given an apparatus to take home. An applicator with a diameter of 9 cm is used. The treatment will be carried out in the morning and evening for 15 minutes each in supine position on a sofa. In accordance with the technique of classical manual lymphatic drainage, stroking and circular movements in the upper and lower leg and the inguinal area take place in a fixed order.
  Other Names: electrostatic fields; electrotherapy
  Arms: Deep Oscillation (DO) self treatment

SUMMARY:
The purpose of this study is to evaluate the effects of Deep Oscillation (DO) self-treatment on recovery after fatiguing soccer training. We investigate deep oscillation (DO) self treatment as a measure to promote regeneration, hypothesizing that DO leads to an accelerated recovery within the first 48h after fatiguing training with positive effect on the maximum strength, rated perceived exertion, creatinkinase (CK) values and DOMS compared to no treatment after an .

DETAILED DESCRIPTION:
Recovery time between in association football (soccer) often is not long enough to completely restore. Insufficient recovery can result in a reduced performance and suboptimal development in the training process and a higher risk for injuries. The purpose of this study is to evaluate the effects of Deep Oscillation (DO) self-treatment on recovery after fatiguing soccer training. Deep Oscillation is a unique method which is characterized by an alternating electrostatic which results in a deep resonance vibration of patients tissue.

Methods: In a randomized crossover study design including 10 soccer players of the 5th german devision the following parameters will be evaluated directly before and 48h after an fatiguing soccer specific exercise: Maximum isokinetic strength of the leg and hip extensors and flexors (Con-Trex® Leg Press, Physiomed, Germany), rating of perceived exertion (RPE) during isokinetic testing (Borg scale 6-20) and creatine kinase (CK) serum levels. Delayed Onset Muscle Soreness (DOMS; visual analogue scale 1-10) will be recorded 24 and 48h post-exercise. At random half of the group will perform a DO self-treatment twice daily (4 applications) for 15 minutes each, whereas the other half gets no intervention. 4 weeks later in a cross-over design the same procedure will be conducted again.

ELIGIBILITY:
Inclusion Criteria:

* active soccer player in of the 5th devision

Exclusion Criteria:

* health problems
* medication with impact on the endpoints

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2018-01-24 (Actual); Study Completion 2018-02-22 (Actual)

PRIMARY OUTCOMES:
Isokinetic maximum leg strength | prae fatiguing exercise and 48hours post
  Maximum isokinetic strength of the leg- extensors and flexors is tested using a ConTrex isokinetic leg press (Physiomed, Laipers-dorf, Germany).

SECONDARY OUTCOMES:
Rating of perceived exertion (RPE) | during isokinetic testing prae fatiguing exercise and 48hours post
  Rating of perceived exertion (RPE) is obtained immediately after the maximum strength test, using Borg´s 20-point scale.
Creatine kinase (CK) | prae fatiguing exercise and 48hours post
  Creatine kinase (CK) level is analysed out of the serum using the Beckmann Coulter Inc. device (Brea, USA).
Delayed Onset Muscle Soreness (DOMS) | 24hours and 48hours postexercise
  Self reported Delayed Onset Muscle Soreness (DOMS) in the lower extremity on the day after the training and the day after using a visual analogue scale (VAS) from 1 (no muscle soreness) to 10 (maximum muscle soreness) .

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Medical Physics, University Erlangen-Nurnberg, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] von Stengel S, Teschler M, Weissenfels A, Willert S, Kemmler W. Effect of deep oscillation as a recovery method after fatiguing soccer training: A randomized cross-over study. J Exerc Sci Fit. 2018 Dec;16(3):112-117. doi: 10.1016/j.jesf.2018.10.004. Epub 2018 Oct 16. PMID 30662504